CLINICAL TRIAL: NCT06533124
Title: Parameters of Cardiac Indices on the Ultrasonic Cardiac Output Monitor As Potential Indicators for Predicting the Achievement of Ultrafiltration Endpoint for Acute Heart Failure Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Tong Ren Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2019-072-01
Record Dates: First submitted 2024-07-29; First posted 2024-08-01 (Actual); Last update posted 2024-08-01 (Actual); Status verified 2024-07

CONDITIONS: Acute Heart Failure
Keywords: Ultrasonic cardiac output monitor (USCOM); Acute heart failure; Brain natriuretic peptide; Ultrafiltration; Echocardiography

STUDY DESIGN:
Intervention Model Description: Patients were randomly assigned in a 1:1 ratio, with one group receiving UF treatment alone and the other receiving UF treatment plus USCOM monitoring. The allocation of study participants was processed through an interactive web response system with a non-stratified permutated block size. Treating clinicians were unaware of patients' group assignments; there were a total of 40 patients.
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- USCOM + ultrafiltration group-experimental group (Experimental): In the USCOM + ultrafiltration group, cardiac output was monitored using a non-invasive ultrasonic cardiac output monitor, which employed transaortic or transpulmonary Doppler flow tracing and estimated the valve area using a patient's height to estimate their cardiac output. The monitored parameters include, SV index (SVI), SV variation (SVV), cardiac output (CO), cardiac index (CI), inotropy (INO), systemic vascular resistance index (SVRI), systemic vascular resistance (SVR), flow time corrected (FTC) and velocity time integral (VTI) .
  Interventions: Device: The ultrasonic cardiac output monitor 1A system (USCOM Ltd., Sydney, Australia) is a non-invasive Doppler stroke volume (SV) technique derived from echocardiography.
- ultrafiltration group-control group (No Intervention): Patients who met the criteria for ultrafiltration were treated with conventional ultrafiltration.

INTERVENTIONS:
Device: The ultrasonic cardiac output monitor 1A system (USCOM Ltd., Sydney, Australia) is a non-invasive Doppler stroke volume (SV) technique derived from echocardiography. — In the USCOM + ultrafiltration group, cardiac output was monitored using a non-invasive ultrasonic cardiac output monitor, which employed transaortic or transpulmonary Doppler flow tracing and estimated the valve area using a patient's height to estimate their cardiac output. The monitored parameters include, SV index (SVI), SV variation (SVV), cardiac output (CO), cardiac index (CI), inotropy (INO), systemic vascular resistance index (SVRI), systemic vascular resistance (SVR), flow time corrected (FTC) and velocity time integral (VTI) .
  Arms: USCOM + ultrafiltration group-experimental group

SUMMARY:
Background: The feasibility of the ultrasonic cardiac output monitor (USCOM)applying for determining ultrafiltration (UF) endpoints during acute heart failure (AHF) treatments was evaluated.

Methods: AHF patients were randomly assigned to UF (U, N=20) and USCOM+UF (UU, N=20) groups. The primary endpoint was differences in the hemodynamics of patients receiving UF alone or UF+USCOM. A prediction model was established.

DETAILED DESCRIPTION:
This study was based on the ACC/AHA/HFSA guidelines for the management of heart failure and involved 40 patients diagnosed with acute decompensated heart failure (ADHF) from January 2022 to July 2023. Patients were randomly assigned to UF (U, N = 20) and USCOM + UF (UU, N = 20) groups.

The inclusion criteria were: (1) Age ≥ 18 years; (2) Male or non-pregnant female patients; (3) Fluid overload manifested by at least two of the following: a) Pitting edema ≥ 2+ of the lower extremities; b) Moist rales in the lungs; c) Jugular venous distention > 10 cm; d) Pulmonary edema or pleural effusion on chest x-ray; e) Paroxysmal nocturnal dyspnea or ≥ two-pillow orthopnea; f) Congestive hepatomegaly or ascites; e) B-type natriuretic peptide (BNP) > 400 pg/mL.

The exclusion criteria were: (1) Hematocrit > 45%; (2) Systolic blood pressure ≤ 90 mmHg and poor peripheral circulation; (3) Contraindications to heparin anticoagulation;(4) Renal insufficiency with a Scr ≥ 3.0 mg/dl or planned renal replacement therapies; (5) Acute coronary syndromes; (6) Life-threatening organ dysfunction caused by a dysregulated host response to infection; (7) Active myocarditis; (8) patients with heart failure attributed to restrictive or hypertrophic cardiomyopathy or uncorrected valvular stenotic disease; (9) infection; (10) malignancies; (11) systemic immune disease; (12) unwillingness to cooperate; (13) withdrawal from the study or death. The study adhered to the principles of the Declaration of Helsinki and the protocols were approved by the Institutional Review Board of our hospital (2019-072-01). Informed consent was obtained from all enrolled patients.

Randomization:

Patients were randomly assigned in a 1:1 ratio, with one group receiving UF treatment alone and the other receiving UF treatment plus USCOM monitoring. The allocation of study participants was processed through an interactive web response system with a non-stratified permutated block size. Treating clinicians were unaware of patients' group assignments; there were a total of 40 patients.

The operator steps of USCOM The operation of USCOM only requires placing the probe in the patient's pulmonary artery window or aortic window for monitoring. In pulmonary artery window monitoring, the probe is positioned beside the right sternal border or upper abdomen to assess blood flow in the pulmonary artery, thereby monitoring pulmonary circulation and right heart function. For aortic window monitoring, the probe is placed at the sternal notch or subclavian fossa (same as the pulmonary artery window), and measurements are taken through the aorta to assess systemic circulation, primarily monitoring left ventricular output. In this study, only one skilled operator monitored all UU group patients.

Assessments Patients were assessed at baseline and throughout the period of treatment. The documented variables were medical history, physical examination data, echocardiography, laboratory blood test monitoring (continuous), including the total UF volume, body weight, patient symptoms, body position, transcutaneous oxygen saturation, degree of edema, leg circumference, abdominal circumference, input-output balance and other variables for 7 days. Adverse events (AEs) were assessed and documented by clinicians within 24 h.

In the USCOM plus UF group, cardiac output was monitored using a non-invasive ultrasonic cardiac output monitor, which employed transaortic or transpulmonary Doppler flow tracing and estimated the valve area using a patient's height to estimate their cardiac output. The monitored parameters included the SV index (SVI), SV variation (SVV), cardiac output (CO), cardiac index (CI), inotropy (INO), systemic vascular resistance index (SVRI), systemic vascular resistance (SVR), flow time corrected (FTC) and the velocity time integral (VTI) USCOM. Thresholds of a 30% or 50% reduction in BNP relative to baseline were set as criteria for reaching the UF endpoint.

Endpoints The primary endpoint was differences in the hemodynamics of patients in the UF alone and UF plus USCOM groups during UF, monitored at 1, 2, 3, 4 and 7 days. The secondary endpoints were the identification of one or more indicators on the USCOM monitor that could predict the endpoint of UF. Additionally, the study assessed the economic benefits between the two groups.

Statistical analysis All analyses and calculations of sample size were performed using SPSS. Student's t-test or analysis of variance (ANOVA) was used to look for differences in continuous regularly distributed variables, and the Kruskal-Wallis test was employed to determine whether there were significant group differences. The findings are presented as the mean ± SD. A Mann-Whitney U test or Wilcoxon rank sum test was used for continuous variables that were not normally distributed, and the results are reported as median (Q1, Q3). To assess potential differences between categorical variables, a χ² test or Fisher's exact test was used for analysis. P-values < 0.05 were deemed to be significant.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Male or non-pregnant female patients.
* Fluid overload manifested by at least two of the following:

  1. Pitting edema ≥ 2+ of the lower extremities
  2. Moist rales in the lungs
  3. Jugular venous distention > 10 cm
  4. Pulmonary edema or pleural effusion on chest x-ray
  5. Paroxysmal nocturnal dyspnea or ≥ two-pillow orthopnea
  6. Congestive hepatomegaly or ascites
  7. B-type natriuretic peptide (BNP) > 400 pg/mL

Exclusion Criteria:

* Hematocrit > 45%.
* Systolic blood pressure ≤ 90 mmHg and poor peripheral circulation.
* Contraindications to heparin anticoagulation.
* Renal insufficiency with a Scr ≥ 3.0 mg/dl or planned renal replacement therapies.
* Acute coronary syndromes.
* Life-threatening organ dysfunction caused by a dysregulated host response to infection.
* Active myocarditis.
* patients with heart failure attributed to restrictive or hypertrophic cardiomyopathy or uncorrected valvular stenotic disease.
* infection.
* malignancies.
* systemic immune disease.
* unwillingness to cooperate.
* withdrawal from the study or death.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2022-01-05 (Actual); Primary Completion 2023-07-05 (Actual); Study Completion 2023-08-01 (Actual)

PRIMARY OUTCOMES:
Cardiac output was monitored using a non-invasive ultrasonic cardiac output monitor, which employed transaortic or transpulmonary Doppler flow tracing and estimated the valve area using a patient's height to estimate their cardiac output. | One week
  SVV, systemic vascular variation, unit of mesure:%
Cardiac output was monitored using a non-invasive ultrasonic cardiac output monitor, which employed transaortic or transpulmonary Doppler flow tracing and estimated the valve area using a patient's height to estimate their cardiac output. | One week
  SVI, systemic vascular index , unit of mesure: ml/m2
Cardiac output was monitored using a non-invasive ultrasonic cardiac output monitor, which employed transaortic or transpulmonary Doppler flow tracing and estimated the valve area using a patient's height to estimate their cardiac output. | One week
  CI, cardiac index, unit of measure: l/min/m2.
Cardiac output was monitored using a non-invasive ultrasonic cardiac output monitor, which employed transaortic or transpulmonary Doppler flow tracing and estimated the valve area using a patient's height to estimate their cardiac output. | One week
  INO, inotropy, unit of measure: w/m2
Cardiac output was monitored using a non-invasive ultrasonic cardiac output monitor, which employed transaortic or transpulmonary Doppler flow tracing and estimated the valve area using a patient's height to estimate their cardiac output. | One week
  CO, cardiac output, unit of measure: l/min.
Cardiac output was monitored using a non-invasive ultrasonic cardiac output monitor, which employed transaortic or transpulmonary Doppler flow tracing and estimated the valve area using a patient's height to estimate their cardiac output. | One week
  SVRI, systemic vascular resistance index, unit of measure: ds cm-5m2.
Cardiac output was monitored using a non-invasive ultrasonic cardiac output monitor, which employed transaortic or transpulmonary Doppler flow tracing and estimated the valve area using a patient's height to estimate their cardiac output. | One week
  SVR, systemic vascular resistance index, unit of measure: ds cm-5.
Cardiac output was monitored using a non-invasive ultrasonic cardiac output monitor, which employed transaortic or transpulmonary Doppler flow tracing and estimated the valve area using a patient's height to estimate their cardiac output. | One week
  FTC, flow time corrected, unit of measure: ms.
Cardiac output was monitored using a non-invasive ultrasonic cardiac output monitor, which employed transaortic or transpulmonary Doppler flow tracing and estimated the valve area using a patient's height to estimate their cardiac output. | One week
  VTI, velocity time integral, unit of measure: cm.
Brain natriuretic peptide | One week
  BNP, Brain natriuretic peptide, unit of measure: pg/ml.

CONTACTS AND LOCATIONS:
Locations (1):
- ShanghaiTongren Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Li Y, Chen J, Bian J, Chen F, Wan Q, Yuan F. Cardiac Indices Parameters on the Ultrasonic Cardiac Output Monitor as Potential Indicators to Predict the Ultrafiltration Endpoint Success in Acute Heart Failure Treatment. Rev Cardiovasc Med. 2025 May 22;26(5):27100. doi: 10.31083/RCM27100. eCollection 2025 May. PMID 40475748